CLINICAL TRIAL: NCT01801475
Title: Prevention of Neonatal Abstinence Syndrome
Brief Title: How Pregnant Women and Their Babies Metabolize Ondansetron Compared to a Group of Non-pregnant Women
Acronym: Zofran_PK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David R. Drover, Professor of Anesthesia, Stanford School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1R01HD070795-01A1 (NIH); NAS Aim 1 (Other: Stanford)
Record Dates: First submitted 2013-01-28; First posted 2013-02-28 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Postoperative Nausea
Keywords: Pharmacokinetics of ondansetron in women; Pharmacokinetics of ondansetron in neonates; Term pregnancy; Cesarean section
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pregnant women (Active Comparator): Full term pregnant women scheduled for Cesarean section and will be given Ondansetron as standard-of-care prior to surgery.
  Interventions: Drug: Ondansetron
- Non-pregnant women (Active Comparator): Non-pregnant women scheduled for surgery at Stanford who will be given Ondansetron prior to their surgery as standard-of-care.
  Interventions: Drug: Ondansetron
- Neonates (No Intervention): Babies of the pregnant women enrolled in the study; no ondansetron is given to babies in this "Aim 1" of the study.

INTERVENTIONS:
Drug: Ondansetron — Pregnant & non-pregnant women will receive either 4mg or 8mg of Ondansetron (IV) once prior to surgical procedure (open-label). Women are in the study for 8 hours. Babies of pregnant women are not given Ondansetron but are in the study for 24-48 hours.
  Other Names: Zofran
  Arms: Non-pregnant women; Pregnant women

SUMMARY:
This is called "Aim 1" of the investigators' NIH grant. Ondansetron (Zofran) is a safe and effective drug used in pregnant women to prevent nausea but the investigators do not know what effect pregnancy may have on the metabolism of Zofran in pregnant women or their babies. Therefore the investigators will enroll approximately 40 pregnant women and their babies and draw blood samples from the mother, the baby and the cord, to determine how much Zofran is in each sample of blood (called the pharmacokinetics or PK of Zofran). The pregnant women will receive Zofran, as a standard-of-care drug, for their scheduled Cesarean Section.

The investigators will also enroll about 20 non-pregnant women undergoing surgery who will receive Zofran as standard-of-care during surgery. In both the pregnant & the non-pregnant women, the investigators will draw blood samples at the same time points based on number of minutes from the time the Zofran is given. The blood data (PK of Zofran) will help the investigators move into Aim 2 of the study, which will be done in pregnant, narcotic-addicted mothers and their babies who are born addicted to narcotics. Aim 2 will be listed separately as it will be an interventional study.

DETAILED DESCRIPTION:
This phase of the study is Aim 1 and it will lead to Aim 2, which specifically will address the Prevention of Neonatal Abstinence Syndrome (NAS).

NAS is a constellation of narcotic drug withdrawal symptoms that develops in 42-94% of the infants born to narcotic dependent mothers. This severe syndrome, of which there are no preventative treatments, can result in prolonged hospitalization, some of which may be in the neonatal intensive care unit (NICU). The investigators have shown that ondansetron can eliminate or alleviate the symptoms of narcotic drug withdrawal in experimental studies in mice and in humans. Based upon these results, it is quite possible that ondansetron administration to pregnant narcotic-using mothers just prior to delivery, followed by a 3-day period of ondansetron administration to the neonate, could reduce the incidence or severity of NAS symptoms.

AIM 1 is a pharmacokinetic (PK) study of intravenous (IV) ondansetron in three different groups of participants: Study Group #1 = non-pregnant women undergoing surgery; Study Group #2 = pregnant women scheduled for cesarean section delivery; Study Group #3 = viable, full term, singleton neonates born to study group #2 mothers. Group #1 will be given IV ondansetron prior to their surgery and up to 5 PK blood samples will be drawn from an indwelling IV line or by IV stick. The PK samples will be 2-5 ml each and will be drawn at baseline (prior to ondansetron) and then at 7, 15, and 40 min and 8 hours after the ondansetron. Group #2 will be given IV ondansetron prior to their cesarean section and up to 6 PK blood samples will be drawn from an indwelling IV line or by IV stick. The PK samples will be 2-5 ml each and will be drawn at baseline, 7, 15, 40 min and prior to delivery and 8 hours after the ondansetron is given. The Group #3 neonates will provide a section of the umbilical cord from which arterial and venous blood samples will be drawn (this section of cord would normally be thrown out and the parents are consenting to allow the Investigators to take these two samples). Each time the baby has a "Standard-of-Care" lab test ordered by heel stick or needle stick, the investigators will obtain a few drops of blood to place on the special research filter paper to determine how much ondansetron is in the baby's blood. If the parents will allow any extra heel sticks, the Investigators will try to obtain 1-2 samples of blood in the first 6 hours of life. If the parents only want their baby's blood taken at the standard-of-care lab draws, then the first scheduled lab draw is at 24 hours of life for the newborn screening which is a mandated by state law. All blood samples taken for this study are being processed by the investigator, not the Stanford Lab. Also, the investigators are doing the PK analysis of the dried blood spots on the filter paper and the analysis of the frozen plasma samples.

Aim 2 of this NIH grant will be entered separately into ClinicalTrials.gov. It will be a multi-center, randomized, double-blind, placebo-controlled trial to determine whether ondansetron treatment will reduce the incidence or severity of NAS in babies born to narcotic-using mothers.

ELIGIBILITY:
Inclusion Criteria:

For Non-pregnant Females (Group #1)

1. Age 18-45 yrs inclusive
2. Generally healthy
3. Undergoing any scheduled surgical procedure deemed suitable by the Investigator MD
4. Planned to receive the drug Ondansetron for the surgery
5. Able and willing to sign the informed consent

For Pregnant Females (Group #2)

1. Age 18-45 yrs inclusive
2. Term pregnancy (37 weeks through 41 wks + 6 days)
3. Generally healthy (not morbidly obese)
4. Undergoing a planned C-section or by an unplanned, non-urgent C-section
5. Planned to receive the drug Ondansetron for the surgery
6. Single birth
7. Able and willing to sign the informed consent for herself & the baby

For the Neonatal Participant (Group #3)

1. Male or female
2. Viable birth
3. Gestational age of 37 weeks through 41 weeks + 6 days
4. Mother gave written consent for baby to participate

Exclusion Criteria:

1. Medical condition that would effect the metabolism of ondansetron
2. Known allergy to ondansetron
3. Use of medications in the last 48 hours, by the pregnant or non-pregnant subjects, that might induce or inhibit the metabolism of ondansetron (such as CYP3A4 inhibitors or inducers)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Drover, MD, Principal Investigator — Stanford University School of Medicine, Department of Anesthesia
Locations (1):
- Lucile Packard Children's Hospital & Stanford Hospital, Palo Alto, California, United States

REFERENCES:
- [Result] Elkomy MH, Sultan P, Carvalho B, Peltz G, Wu M, Clavijo C, Galinkin JL, Drover DR. Ondansetron pharmacokinetics in pregnant women and neonates: towards a new treatment for neonatal abstinence syndrome. Clin Pharmacol Ther. 2015 Feb;97(2):167-76. doi: 10.1002/cpt.5. Epub 2014 Dec 4. PMID 25670522

RESULTS

PARTICIPANT FLOW:
Groups:
- Ondansetron 4 mg IV - Pregnant: Ondansetron 4 mg was given intravenously prior to delivery of the infant.
- Ondansetron 8 mg IV - Pregnant: Ondansetron 8 mg was given intravenously prior to delivery of the infant.
- Non-pregnant Women - 8 mg Ondansetron: As a comparison for pharmacokinetics, a non-pregnant group was enrolled and received ondansetron. 8 mg ondansetron
- Non-pregnant Women - 4 mg Ondansetron: As a comparison for pharmacokinetics, a non-pregnant group was enrolled and received ondansetron. 4 mg ondansetron
- Neonates: The neonates became part of the subject population after birth. They were subsequently sampled for pharmacokinetic samples.
Period: Overall Study
Arm/Group | Ondansetron 4 mg IV - Pregnant | Ondansetron 8 mg IV - Pregnant | Non-pregnant Women - 8 mg Ondansetron | Non-pregnant Women - 4 mg Ondansetron | Neonates
Started | 10 | 30 | 10 | 10 | 40
Completed | 10 | 30 | 10 | 10 | 39
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 3 groups of individual subjects
Groups:
- Pregnant Women: Full term pregnant women scheduled for Cesarean section and will be given Ondansetron as standard-of-care prior to surgery.
  Ondansetron: Pregnant women will receive either 4mg or 8mg of Ondansetron (IV) once prior to surgical procedure (open-label). Women are in the study for 8 hours.
- Non-pregnant Women: Non-pregnant women scheduled for surgery at Stanford who will be given Ondansetron prior to their surgery as standard-of-care.
  Ondansetron: non-pregnant women will receive either 4mg or 8mg of Ondansetron (IV) once prior to surgical procedure (open-label). Women are in the study for 8 hours.
- Neonates: Babies of the pregnant women enrolled in the study; no ondansetron is given to babies in this "Aim 1" of the study. Babies of pregnant women are not given Ondansetron but are in the study for 24-48 hours.
- Total: Total of all reporting groups
Arm/Group | Pregnant Women | Non-pregnant Women | Neonates | Total
Number analyzed (Participants) | 40 | 20 | 39 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] — Neonates were in their first day of life thus their age in years is a very small number.
  A mean of all participants is not relevant for this reason.
  years | 33 (5.2) | 37.7 (5.7) | 0.003 (0.001) | 35 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 20 | 20 | 80
  Male | 0 | 0 | 19 | 19
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 39 | 99

OUTCOME MEASURES:

1. Primary Outcome: Volume of Distribution Estimated Pharmacokinetic Parameter
Description: This is an estimated pharmacokinetic parameter as calculated by NONMEM.
Time Frame: 8 hours for women; 48 hours for neonate.
Population: All subjects but not possible for neonates
Measure: Mean (95% Confidence Interval); unit: Liters
Groups:
- Women - Pregnant/Non-pregnant: Ondansetron 4 mg or 8mg was given intravenously prior to delivery of her baby in pregnant women and was given to age similar women in the non-pregnant group.
Arm/Group | Women - Pregnant/Non-pregnant | Neonates
Number analyzed (Participants) | 60 | 39
Liters | 27.9 [18.5 to 37.3] | NA [NA to NA] — Sampling schedule and dose route would not allow mathematical estimation.
Statistical Analysis 1: Comparison: Women - Pregnant/Non-pregnant; The nonlinear mixed-effects modeling software program NONMEM (version VII; Icon Development Solutions, Ellicott City, MD) was used to estimate the pharmacokinetic parameters. The first-order conditional estimation (FOCE) with η-ε interaction was used for the estimation process. Volume and clearance in this model is computed as a mean of the study population (pregnant and non-pregnant women) with a log-normal distribution in the population; Test type: Superiority or Other; p < 0.05, Chi-squared

2. Primary Outcome: Metabolic Clearance of Ondasetron
Description: This is a mathematical estimation of the clearance for ondasetron as calculated by NONMEM.
Time Frame: 8 hours for women; 48 hours for neonate.
Population: All patient data was used in the estimation process.
Measure: Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Women - Pregnant/Non-pregnant | Neonates
Number analyzed (Participants) | 60 | 39
L/hr | 21.8 [18.9 to 24.6] | NA [NA to NA] — The lack of a direct dose of ondansetron and sufficient sampling made it incorrect to estimate a clearance in the neonate.
Statistical Analysis 1: Comparison: Women - Pregnant/Non-pregnant; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: From time of administration of ondansetron until last sample of blood for pharmacokinetic analysis at 8 hours.
Arm/Group | Ondansetron 4 mg IV - Pregnant | Ondansetron 8 mg IV - Pregnant | Non-pregnant Women - 8 mg Ondansetron | Non-pregnant Women - 4 mg Ondansetron | Neonates
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/30 | 0/10 | 0/10 | 0/40
Other Adverse Events (participants affected / at risk) | 0/10 | 0/30 | 0/10 | 0/10 | 0/40

LIMITATIONS AND CAVEATS:
Since the neonate was not given a dose of study medication (ondansetron) directly it was not possible to estimate the volume of distribution in the neonate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No